CLINICAL TRIAL: NCT05750212
Title: Musculoskeletal and Pelvic Floor Health in Female Chronic Overlapping Pelvic Pain Conditions (The MSK-PELVIC Study)
Brief Title: Musculoskeletal and Pelvic Floor Health in Female Chronic Overlapping Pelvic Pain Conditions
Status: Recruiting | Type: Observational
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Colleen M. Fitzgerald, MD, MS, Principal Investigator, Loyola University
Other Study IDs: 213778
Record Dates: First submitted 2023-01-20; First posted 2023-03-01 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pelvic Pain Syndrome
MeSH Terms: interventions — Electromyography; Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Cases are adult female patients with a diagnosis of pelvic floor disorder.
  Interventions: Diagnostic Test: Tone; Diagnostic Test: Tenderness; Diagnostic Test: Contraction; Diagnostic Test: Relaxation; Diagnostic Test: Electromyography; Diagnostic Test: Transperineal; Diagnostic Test: Pressure
- Controls: Controls are adult female patients sampled from an outpatient primary care center
  Interventions: Diagnostic Test: Tone; Diagnostic Test: Tenderness; Diagnostic Test: Contraction; Diagnostic Test: Relaxation; Diagnostic Test: Electromyography; Diagnostic Test: Transperineal; Diagnostic Test: Pressure

INTERVENTIONS:
Diagnostic Test: Tone — Tone is a binary measurement of the pelvic floor muscle on physical examination
Diagnostic Test: Tenderness — Tenderness is a binary measurement of the pelvic floor muscle on physical examination
Diagnostic Test: Contraction — Contraction is a binary measurement of the pelvic floor muscle on physical examination
Diagnostic Test: Relaxation — Relaxation is a binary measurement of the pelvic floor muscle on physical examination
Diagnostic Test: Electromyography — Electromyography is a measurement of the pelvic floor muscle in microvolts
Diagnostic Test: Transperineal — Transperineal measurements (in millimeters) of the pelvic floor muscle using an ultrasound
Diagnostic Test: Pressure — Pressure measurements (in millimeters) of the pelvic floor muscle using an algometer

SUMMARY:
The purpose of this study is to learn about nerve function and pelvic muscle function. To do this we will compare the pelvic nerve and muscle function of women with chronic pelvic pain to those who do not have chronic pelvic pain. Understanding the pain may lead to better treatments in the future.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) may affect up to a quarter of all women. Traditionally, CPP has been thought to be driven by visceral pain mechanisms such as Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS), Irritable bowel syndrome (IBS) and endometriosis. It is also established that these visceral pain conditions overlap with vulvodynia, fibromyalgia, depression, and anxiety. More recently, underlying pelvic floor myofascial (PFMP) and dyssynergia have been identified as additional overlapping CPP conditions. Prior work suggests PFMP may be a viscero-somatic response, however, PFMP as a compensatory consequence of other regional musculoskeletal (MSK) conditions has also been proposed. Indeed, across their lifespan, women face higher risks than men for a plethora of MSK injuries and chronic MSK conditions, including an increased prevalence of sports-related injuries, joint hypermobility, fibromyalgia, osteoarthritic conditions (post-menopause), and osteoporosis/osteoporosis-associated fractures. These elevated risks are thought to be due to the unique anatomic (structural), biomechanical, and hormonal factors that can be attributed to the physiologic process of pregnancy and aging. The current application aims to address the significant knowledge gap regarding the limited understanding of the neuromuscular function of the PFM in CPP as well as the role of overlapping MSK conditions and MSK health that may be influencing PFM response. The short-term goal is to examine PFM biomechanics by identifying the most precise muscle measures in women with CPP of various overlapping diagnoses compared to asymptomatic controls, along with assessing overall MSK health/physical activity. The long-term goal is to determine MSK pelvic pain mechanisms that will inform clinically relevant classification, develop evidence-based non-pharmacologic (physical therapy/exercise) treatments for women with CPP, and advance research tools in the area of PFM function and CPP as it relates to overall MSK health. Our innovative strategy combines neuromuscular measures using novel devices and validated measures in evaluating CPP, MSK health, and physical activity. Our central hypothesis is that women with CPP will demonstrate quantifiable PFM abnormalities and clinical MSK characteristics that differ from asymptomatic controls. The results from this study will have a significant public health impact with contributions of rigorous objective and comprehensive PFM and MSK methods, which will be suitable for future NIH clinical research networks/trials, to evaluate and assess the MSK contribution and potential treatment outcomes in women with CPP.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 21 to 80 years
* Symptoms of CPP as defined by the American College of Obstetrics & Gynecology (ACOG) for more than 6 months
* At least two of seven overlapping CPP diagnosis (i.e., IC/PBS, IBS, Endometriosis, Vulvodynia, PN, FM, PFMP)
* An average CPP pain score of at least three on a 10 point pain scale

Exclusion Criteria:

* Current or history of GI or GU pelvic cancer
* Current pelvic infection (e.g., a UTI or vaginal infection)
* Current or imminent planned pregnancy or recent delivery in the last 6 months
* Abdominal or pelvic surgery in the last 36 months.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are selected from a tertiary medical care center
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-09-24 (Estimated); Study Completion 2025-10-24 (Estimated)

PRIMARY OUTCOMES:
Difference in two receiver operating characteristic curves | 0 Days
  The delta value between two diagnostic accuracy statistics (c-statistics) will be reported with its 95% confidence interval and significance value (p-value).

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Fitzgerald, MD, Principal Investigator — Loyola Medical Center
Locations (1):
- Loyola Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahangari A. Prevalence of chronic pelvic pain among women: an updated review. Pain Physician. 2014 Mar-Apr;17(2):E141-7. PMID 24658485
- [Background] Bullones Rodriguez MA, Afari N, Buchwald DS; National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Urological Chronic Pelvic Pain. Evidence for overlap between urological and nonurological unexplained clinical conditions. J Urol. 2013 Jan;189(1 Suppl):S66-74. doi: 10.1016/j.juro.2012.11.019. PMID 23234637
- [Background] Harte SE, Schrepf A, Gallop R, Kruger GH, Lai HHH, Sutcliffe S, Halvorson M, Ichesco E, Naliboff BD, Afari N, Harris RE, Farrar JT, Tu F, Landis JR, Clauw DJ; MAPP Research Network. Quantitative assessment of nonpelvic pressure pain sensitivity in urologic chronic pelvic pain syndrome: a MAPP Research Network study. Pain. 2019 Jun;160(6):1270-1280. doi: 10.1097/j.pain.0000000000001505. PMID 31050659
- [Background] Liu A, Chedid V, Wang XJ, Vijayvargiya P, Camilleri M. Clinical presentation and characteristics of pelvic floor myofascial pain in patients presenting with constipation. Neurogastroenterol Motil. 2020 Jul;32(7):e13845. doi: 10.1111/nmo.13845. Epub 2020 Apr 13. PMID 32281205
- [Background] Lamvu G, Carrillo J, Witzeman K, Alappattu M. Musculoskeletal Considerations in Female Patients with Chronic Pelvic Pain. Semin Reprod Med. 2018 Mar;36(2):107-115. doi: 10.1055/s-0038-1676085. Epub 2018 Dec 19. PMID 30566976
- [Background] Ye AL, Adams W, Westbay LC, Fitzgerald CM. Evaluating Disability-Related Quality of Life in Women With Chronic Pelvic Pain. Female Pelvic Med Reconstr Surg. 2020 Aug;26(8):508-513. doi: 10.1097/SPV.0000000000000771. PMID 31425373
- [Background] Hootman JM, Dick R, Agel J. Epidemiology of collegiate injuries for 15 sports: summary and recommendations for injury prevention initiatives. J Athl Train. 2007 Apr-Jun;42(2):311-9. PMID 17710181
- [Background] Wentz L, Liu PY, Haymes E, Ilich JZ. Females have a greater incidence of stress fractures than males in both military and athletic populations: a systemic review. Mil Med. 2011 Apr;176(4):420-30. doi: 10.7205/milmed-d-10-00322. PMID 21539165
- [Background] Agel J, Arendt EA, Bershadsky B. Anterior cruciate ligament injury in national collegiate athletic association basketball and soccer: a 13-year review. Am J Sports Med. 2005 Apr;33(4):524-30. doi: 10.1177/0363546504269937. Epub 2005 Feb 8. PMID 15722283
- [Background] Gwinn DE, Wilckens JH, McDevitt ER, Ross G, Kao TC. The relative incidence of anterior cruciate ligament injury in men and women at the United States Naval Academy. Am J Sports Med. 2000 Jan-Feb;28(1):98-102. doi: 10.1177/03635465000280012901. PMID 10653551
- [Background] Arendt E, Dick R. Knee injury patterns among men and women in collegiate basketball and soccer. NCAA data and review of literature. Am J Sports Med. 1995 Nov-Dec;23(6):694-701. doi: 10.1177/036354659502300611. PMID 8600737
- [Background] O'Connor KL, Baker MM, Dalton SL, Dompier TP, Broglio SP, Kerr ZY. Epidemiology of Sport-Related Concussions in High School Athletes: National Athletic Treatment, Injury and Outcomes Network (NATION), 2011-2012 Through 2013-2014. J Athl Train. 2017 Mar;52(3):175-185. doi: 10.4085/1062-6050-52.1.15. PMID 28387555
- [Background] Zuckerman SL, Kerr ZY, Yengo-Kahn A, Wasserman E, Covassin T, Solomon GS. Epidemiology of Sports-Related Concussion in NCAA Athletes From 2009-2010 to 2013-2014: Incidence, Recurrence, and Mechanisms. Am J Sports Med. 2015 Nov;43(11):2654-62. doi: 10.1177/0363546515599634. Epub 2015 Sep 1. PMID 26330572
- [Background] Smith BE, Selfe J, Thacker D, Hendrick P, Bateman M, Moffatt F, Rathleff MS, Smith TO, Logan P. Incidence and prevalence of patellofemoral pain: A systematic review and meta-analysis. PLoS One. 2018 Jan 11;13(1):e0190892. doi: 10.1371/journal.pone.0190892. eCollection 2018. PMID 29324820
- [Background] Hunt KJ, Hurwit D, Robell K, Gatewood C, Botser IB, Matheson G. Incidence and Epidemiology of Foot and Ankle Injuries in Elite Collegiate Athletes. Am J Sports Med. 2017 Feb;45(2):426-433. doi: 10.1177/0363546516666815. Epub 2016 Nov 2. PMID 27802962
- [Background] Russek LN, Errico DM. Prevalence, injury rate and, symptom frequency in generalized joint laxity and joint hypermobility syndrome in a "healthy" college population. Clin Rheumatol. 2016 Apr;35(4):1029-39. doi: 10.1007/s10067-015-2951-9. Epub 2015 May 1. PMID 25930211
- [Background] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367
- [Background] Prieto-Alhambra D, Judge A, Javaid MK, Cooper C, Diez-Perez A, Arden NK. Incidence and risk factors for clinically diagnosed knee, hip and hand osteoarthritis: influences of age, gender and osteoarthritis affecting other joints. Ann Rheum Dis. 2014 Sep;73(9):1659-64. doi: 10.1136/annrheumdis-2013-203355. Epub 2013 Jun 6. PMID 23744977
- [Background] D'Ambrosia RD. Epidemiology of osteoarthritis. Orthopedics. 2005 Feb;28(2 Suppl):s201-5. doi: 10.3928/0147-7447-20050202-04. PMID 15747607
- [Background] Compston JE, McClung MR, Leslie WD. Osteoporosis. Lancet. 2019 Jan 26;393(10169):364-376. doi: 10.1016/S0140-6736(18)32112-3. PMID 30696576
- [Background] Dugan SA, Gabriel KP, Lange-Maia BS, Karvonen-Gutierrez C. Physical Activity and Physical Function: Moving and Aging. Obstet Gynecol Clin North Am. 2018 Dec;45(4):723-736. doi: 10.1016/j.ogc.2018.07.009. Epub 2018 Oct 25. PMID 30401553
- [Background] Dugan SA, Powell LH, Kravitz HM, Everson Rose SA, Karavolos K, Luborsky J. Musculoskeletal pain and menopausal status. Clin J Pain. 2006 May;22(4):325-31. doi: 10.1097/01.ajp.0000208249.07949.d5. PMID 16691084
- [Background] Lange-Maia BS, Karvonen-Gutierrez CA, Kazlauskaite R, Strotmeyer ES, Karavolos K, Appelhans BM, Janssen I, Avery EF, Dugan SA, Kravitz HM. Impact of Chronic Medical Condition Development on Longitudinal Physical Function from Mid- to Early Late-Life: The Study of Women's Health Across the Nation. J Gerontol A Biol Sci Med Sci. 2020 Jun 18;75(7):1411-1417. doi: 10.1093/gerona/glz243. PMID 31732730
- [Background] Pettee Gabriel K, Sternfeld B, Colvin A, Stewart A, Strotmeyer ES, Cauley JA, Dugan S, Karvonen-Gutierrez C. Physical activity trajectories during midlife and subsequent risk of physical functioning decline in late mid-life: The Study of Women's Health Across the Nation (SWAN). Prev Med. 2017 Dec;105:287-294. doi: 10.1016/j.ypmed.2017.10.005. Epub 2017 Oct 5. PMID 28987336
- [Background] Waetjen LE, Crawford SL, Chang PY, Reed BD, Hess R, Avis NE, Harlow SD, Greendale GA, Dugan SA, Gold EB; Study of Women's Health Across the Nation (SWAN). Factors associated with developing vaginal dryness symptoms in women transitioning through menopause: a longitudinal study. Menopause. 2018 Oct;25(10):1094-1104. doi: 10.1097/GME.0000000000001130. PMID 29916947
- [Background] Rurangirwa AA, Gaillard R, Steegers EA, Hofman A, Jaddoe VW. Hemodynamic adaptations in different trimesters among nulliparous and multiparous pregnant women; the Generation R study. Am J Hypertens. 2012 Aug;25(8):892-9. doi: 10.1038/ajh.2012.57. Epub 2012 May 31. PMID 22647784
- [Background] Hill CC, Pickinpaugh J. Physiologic changes in pregnancy. Surg Clin North Am. 2008 Apr;88(2):391-401, vii. doi: 10.1016/j.suc.2007.12.005. PMID 18381119
- [Background] San-Frutos L, Engels V, Zapardiel I, Perez-Medina T, Almagro-Martinez J, Fernandez R, Bajo-Arenas JM. Hemodynamic changes during pregnancy and postpartum: a prospective study using thoracic electrical bioimpedance. J Matern Fetal Neonatal Med. 2011 Nov;24(11):1333-40. doi: 10.3109/14767058.2011.556203. Epub 2011 Feb 22. PMID 21338331
- [Background] Elkus R, Popovich J Jr. Respiratory physiology in pregnancy. Clin Chest Med. 1992 Dec;13(4):555-65. PMID 1478018
- [Background] Knuttgen HG, Emerson K Jr. Physiological response to pregnancy at rest and during exercise. J Appl Physiol. 1974 May;36(5):549-53. doi: 10.1152/jappl.1974.36.5.549. No abstract available. PMID 4826317
- [Background] ACOG Committee Opinion No. 650: Physical Activity and Exercise During Pregnancy and the Postpartum Period. Obstet Gynecol. 2015 Dec;126(6):e135-e142. doi: 10.1097/AOG.0000000000001214. PMID 26595585
- [Background] Heckman JD, Sassard R. Musculoskeletal considerations in pregnancy. J Bone Joint Surg Am. 1994 Nov;76(11):1720-30. doi: 10.2106/00004623-199411000-00018. No abstract available. PMID 7962034
- [Background] FitzGerald MP, Payne CK, Lukacz ES, Yang CC, Peters KM, Chai TC, Nickel JC, Hanno PM, Kreder KJ, Burks DA, Mayer R, Kotarinos R, Fortman C, Allen TM, Fraser L, Mason-Cover M, Furey C, Odabachian L, Sanfield A, Chu J, Huestis K, Tata GE, Dugan N, Sheth H, Bewyer K, Anaeme A, Newton K, Featherstone W, Halle-Podell R, Cen L, Landis JR, Propert KJ, Foster HE Jr, Kusek JW, Nyberg LM; Interstitial Cystitis Collaborative Research Network. Randomized multicenter clinical trial of myofascial physical therapy in women with interstitial cystitis/painful bladder syndrome and pelvic floor tenderness. J Urol. 2012 Jun;187(6):2113-8. doi: 10.1016/j.juro.2012.01.123. Epub 2012 Apr 12. PMID 22503015
- [Background] Halder GE, Scott L, Wyman A, Mora N, Miladinovic B, Bassaly R, Hoyte L. Botox combined with myofascial release physical therapy as a treatment for myofascial pelvic pain. Investig Clin Urol. 2017 Mar;58(2):134-139. doi: 10.4111/icu.2017.58.2.134. Epub 2017 Feb 1. PMID 28261683
- [Background] Bartley J, Han E, Gupta P, Gaines N, Killinger KA, Boura JA, Farrah M, Gilleran J, Sirls LT, Peters KM. Transvaginal Trigger Point Injections Improve Pain Scores in Women with Pelvic Floor Hypertonicity and Pelvic Pain Conditions. Female Pelvic Med Reconstr Surg. 2019 Sep/Oct;25(5):392-396. doi: 10.1097/SPV.0000000000000581. PMID 29621041
- [Background] Carey ET, Till SR, As-Sanie S. Pharmacological Management of Chronic Pelvic Pain in Women. Drugs. 2017 Mar;77(3):285-301. doi: 10.1007/s40265-016-0687-8. PMID 28074359
- [Background] Andrews J, Yunker A, Reynolds WS, Likis FE, Sathe NA, Jerome RN. Noncyclic Chronic Pelvic Pain Therapies for Women: Comparative Effectiveness [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2012 Jan. Report No.: 11(12)-EHC088-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK84586/ PMID 22439157
- [Background] Carter JE. Surgical treatment for chronic pelvic pain. JSLS. 1998 Apr-Jun;2(2):129-39. PMID 9876726
- [Background] AbdelHafeez MA, Reda A, Elnaggar A, El-Zeneiny H, Mokhles JM. Gabapentin for the management of chronic pelvic pain in women. Arch Gynecol Obstet. 2019 Nov;300(5):1271-1277. doi: 10.1007/s00404-019-05272-z. Epub 2019 Aug 21. PMID 31435774
- [Background] Chronic Pelvic Pain: ACOG Practice Bulletin, Number 218. Obstet Gynecol. 2020 Mar;135(3):e98-e109. doi: 10.1097/AOG.0000000000003716. PMID 32080051
- [Background] TAVERNER D, SMIDDY FG. An electromyographic study of the normal function of the external anal sphincter and pelvic diaphragm. Dis Colon Rectum. 1959 Mar-Apr;2(2):153-60. doi: 10.1007/BF02616708. No abstract available. PMID 13652783
- [Background] Sapsford RR, Hodges PW, Richardson CA, Cooper DH, Markwell SJ, Jull GA. Co-activation of the abdominal and pelvic floor muscles during voluntary exercises. Neurourol Urodyn. 2001;20(1):31-42. doi: 10.1002/1520-6777(2001)20:13.0.co;2-p. PMID 11135380
- [Background] Sapsford RR, Richardson CA, Maher CF, Hodges PW. Pelvic floor muscle activity in different sitting postures in continent and incontinent women. Arch Phys Med Rehabil. 2008 Sep;89(9):1741-7. doi: 10.1016/j.apmr.2008.01.029. PMID 18760158
- [Background] Weiss JM. Pelvic floor myofascial trigger points: manual therapy for interstitial cystitis and the urgency-frequency syndrome. J Urol. 2001 Dec;166(6):2226-31. doi: 10.1016/s0022-5347(05)65539-5. PMID 11696740
- [Background] Bassaly R, Tidwell N, Bertolino S, Hoyte L, Downes K, Hart S. Myofascial pain and pelvic floor dysfunction in patients with interstitial cystitis. Int Urogynecol J. 2011 Apr;22(4):413-8. doi: 10.1007/s00192-010-1301-3. Epub 2010 Oct 26. PMID 20976441
- [Background] Tu FF, As-Sanie S, Steege JF. Musculoskeletal causes of chronic pelvic pain: a systematic review of existing therapies: part II. Obstet Gynecol Surv. 2005 Jul;60(7):474-83. doi: 10.1097/01.ogx.0000162246.06900.9f. PMID 15995564
- [Background] Tu FF, As-Sanie S, Steege JF. Prevalence of pelvic musculoskeletal disorders in a female chronic pelvic pain clinic. J Reprod Med. 2006 Mar;51(3):185-9. PMID 16674013
- [Background] Peters KM, Carrico DJ, Diokno AC. Characterization of a clinical cohort of 87 women with interstitial cystitis/painful bladder syndrome. Urology. 2008 Apr;71(4):634-40. doi: 10.1016/j.urology.2007.11.013. PMID 18387392
- [Background] Tu FF, Holt J, Gonzales J, Fitzgerald CM. Physical therapy evaluation of patients with chronic pelvic pain: a controlled study. Am J Obstet Gynecol. 2008 Mar;198(3):272.e1-7. doi: 10.1016/j.ajog.2007.09.002. PMID 18313447
- [Background] Butrick CW. Pelvic floor hypertonic disorders: identification and management. Obstet Gynecol Clin North Am. 2009 Sep;36(3):707-22. doi: 10.1016/j.ogc.2009.08.011. PMID 19932423
- [Background] Fitzgerald CM, Neville CE, Mallinson T, Badillo SA, Hynes CK, Tu FF. Pelvic floor muscle examination in female chronic pelvic pain. J Reprod Med. 2011 Mar-Apr;56(3-4):117-22. PMID 21542528
- [Background] Meister MR, Sutcliffe S, Ghetti C, Chu CM, Spitznagle T, Warren DK, Lowder JL. Development of a standardized, reproducible screening examination for assessment of pelvic floor myofascial pain. Am J Obstet Gynecol. 2019 Mar;220(3):255.e1-255.e9. doi: 10.1016/j.ajog.2018.11.1106. Epub 2018 Dec 7. PMID 30527941
- [Background] Frawley H, Shelly B, Morin M, Bernard S, Bo K, Digesu GA, Dickinson T, Goonewardene S, McClurg D, Rahnama'i MS, Schizas A, Slieker-Ten Hove M, Takahashi S, Voelkl Guevara J. An International Continence Society (ICS) report on the terminology for pelvic floor muscle assessment. Neurourol Urodyn. 2021 Jun;40(5):1217-1260. doi: 10.1002/nau.24658. Epub 2021 Apr 12. PMID 33844342
- [Background] Beales DJ, O'Sullivan PB, Briffa NK. Motor control patterns during an active straight leg raise in chronic pelvic girdle pain subjects. Spine (Phila Pa 1976). 2009 Apr 20;34(9):861-70. doi: 10.1097/BRS.0b013e318198d212. PMID 19531994
- [Background] Glazer HI, Jantos M, Hartmann EH, Swencionis C. Electromyographic comparisons of the pelvic floor in women with dysesthetic vulvodynia and asymptomatic women. J Reprod Med. 1998 Nov;43(11):959-62. PMID 9839264
- [Background] Grape HH, Dedering A, Jonasson AF. Retest reliability of surface electromyography on the pelvic floor muscles. Neurourol Urodyn. 2009;28(5):395-9. doi: 10.1002/nau.20648. PMID 19214991
- [Background] Dias N, Zhang C, Spitznagle T, Lai HH, Zhang Y. High-Density Surface Electromyography Assessment of Pelvic Floor Dysfunction in Women with Interstitial Cystitis/Bladder Pain Syndrome. J Urol. 2020 Dec;204(6):1275-1283. doi: 10.1097/JU.0000000000001237. Epub 2020 Jul 6. PMID 32628100
- [Background] Peschers UM, Gingelmaier A, Jundt K, Leib B, Dimpfl T. Evaluation of pelvic floor muscle strength using four different techniques. Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(1):27-30. doi: 10.1007/s001920170090. PMID 11294527
- [Background] Stuge B, Saetre K, Braekken IH. The association between pelvic floor muscle function and pelvic girdle pain--a matched case control 3D ultrasound study. Man Ther. 2012 Apr;17(2):150-6. doi: 10.1016/j.math.2011.12.004. Epub 2012 Jan 15. PMID 22245422
- [Background] Polpeta NC, Giraldo PC, Juliato CR, Yoshida LP, do Amaral RL, Eleuterio J Jr. Electromyography and vaginal pressure of the pelvic floor muscles in women with recurrent vulvovaginal candidiasis and vulvodynia. J Reprod Med. 2012 Mar-Apr;57(3-4):141-7. PMID 22523874
- [Background] Voorham-van der Zalm PJ, Voorham JC, van den Bos TW, Ouwerkerk TJ, Putter H, Wasser MN, Webb A, DeRuiter MC, Pelger RC. Reliability and differentiation of pelvic floor muscle electromyography measurements in healthy volunteers using a new device: the Multiple Array Probe Leiden (MAPLe). Neurourol Urodyn. 2013 Apr;32(4):341-8. doi: 10.1002/nau.22311. Epub 2012 Sep 12. PMID 22972554
- [Background] Voorham JC, De Wachter S, Van den Bos TWL, Putter H, Lycklama A Nijeholt GA, Voorham-van der Zalm PJ. The effect of EMG biofeedback assisted pelvic floor muscle therapy on symptoms of the overactive bladder syndrome in women: A randomized controlled trial. Neurourol Urodyn. 2017 Sep;36(7):1796-1803. doi: 10.1002/nau.23180. Epub 2016 Nov 21. PMID 27869312
- [Background] Huskisson EC. Measurement of pain. J Rheumatol. 1982 Sep-Oct;9(5):768-9. No abstract available. PMID 6184474
- [Background] Lapin B, Davin S, Stilphen M, Benzel E, Katzan IL. Validation of PROMIS CATs and PROMIS Global Health in an Interdisciplinary Pain Program for Patients With Chronic Low Back Pain. Spine (Phila Pa 1976). 2020 Feb 15;45(4):E227-E235. doi: 10.1097/BRS.0000000000003232. PMID 31513107
- [Background] van den Hoven LH, Gorter KJ, Picavet HS. Measuring musculoskeletal pain by questionnaires: the manikin versus written questions. Eur J Pain. 2010 Mar;14(3):335-8. doi: 10.1016/j.ejpain.2009.06.002. Epub 2009 Aug 20. PMID 19699125
- [Background] Pollard CA. Preliminary validity study of the pain disability index. Percept Mot Skills. 1984 Dec;59(3):974. doi: 10.2466/pms.1984.59.3.974. No abstract available. PMID 6240632
- [Background] Tait RC, Pollard CA, Margolis RB, Duckro PN, Krause SJ. The Pain Disability Index: psychometric and validity data. Arch Phys Med Rehabil. 1987 Jul;68(7):438-41. PMID 3606368
- [Background] Hill JC, Kang S, Benedetto E, Myers H, Blackburn S, Smith S, Dunn KM, Hay E, Rees J, Beard D, Glyn-Jones S, Barker K, Ellis B, Fitzpatrick R, Price A. Development and initial cohort validation of the Arthritis Research UK Musculoskeletal Health Questionnaire (MSK-HQ) for use across musculoskeletal care pathways. BMJ Open. 2016 Aug 5;6(8):e012331. doi: 10.1136/bmjopen-2016-012331. PMID 27496243
- [Background] Rosen RC. Measurement of male and female sexual dysfunction. Curr Psychiatry Rep. 2001 Jun;3(3):182-7. doi: 10.1007/s11920-001-0050-x. PMID 11353580
- [Background] O'Leary MP, Sant GR, Fowler FJ Jr, Whitmore KE, Spolarich-Kroll J. The interstitial cystitis symptom index and problem index. Urology. 1997 May;49(5A Suppl):58-63. doi: 10.1016/s0090-4295(99)80333-1. PMID 9146003
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Background] Jones G, Jenkinson C, Kennedy S. Development of the Short Form Endometriosis Health Profile Questionnaire: the EHP-5. Qual Life Res. 2004 Apr;13(3):695-704. doi: 10.1023/B:QURE.0000021321.48041.0e. PMID 15130031
- [Background] Sullivan MJ, D'Eon JL. Relation between catastrophizing and depression in chronic pain patients. J Abnorm Psychol. 1990 Aug;99(3):260-3. doi: 10.1037//0021-843x.99.3.260. PMID 2145334
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Lin I, Wiles L, Waller R, Goucke R, Nagree Y, Gibberd M, Straker L, Maher CG, O'Sullivan PPB. What does best practice care for musculoskeletal pain look like? Eleven consistent recommendations from high-quality clinical practice guidelines: systematic review. Br J Sports Med. 2020 Jan;54(2):79-86. doi: 10.1136/bjsports-2018-099878. Epub 2019 Mar 2. PMID 30826805
- [Background] Majlesi J, Togay H, Unalan H, Toprak S. The sensitivity and specificity of the Slump and the Straight Leg Raising tests in patients with lumbar disc herniation. J Clin Rheumatol. 2008 Apr;14(2):87-91. doi: 10.1097/RHU.0b013e31816b2f99. PMID 18391677
- [Background] Maitland GD. The slump test: examination and treatment. Aust J Physiother. 1985;31(6):215-9. doi: 10.1016/S0004-9514(14)60634-6. PMID 25026106
- [Background] Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. doi: 10.1007/s00586-008-0602-4. Epub 2008 Feb 8. PMID 18259783
- [Background] Mens JM, Vleeming A, Snijders CJ, Koes BW, Stam HJ. Reliability and validity of the active straight leg raise test in posterior pelvic pain since pregnancy. Spine (Phila Pa 1976). 2001 May 15;26(10):1167-71. doi: 10.1097/00007632-200105150-00015. PMID 11413432
- [Background] Mens JM, Vleeming A, Snijders CJ, Stam HJ, Ginai AZ. The active straight leg raising test and mobility of the pelvic joints. Eur Spine J. 1999;8(6):468-73. doi: 10.1007/s005860050206. PMID 10664304
- [Background] Friedrich J, Brakke R, Akuthota V, Sullivan W. Reliability and Practicality of the Core Score: Four Dynamic Core Stability Tests Performed in a Physician Office Setting. Clin J Sport Med. 2017 Jul;27(4):409-414. doi: 10.1097/JSM.0000000000000366. PMID 28653966
- [Background] Kockum B, Heijne AI. Hop performance and leg muscle power in athletes: Reliability of a test battery. Phys Ther Sport. 2015 Aug;16(3):222-7. doi: 10.1016/j.ptsp.2014.09.002. Epub 2014 Sep 19. PMID 25891995
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Dietz HP. Ultrasound imaging of the pelvic floor. Part I: two-dimensional aspects. Ultrasound Obstet Gynecol. 2004 Jan;23(1):80-92. doi: 10.1002/uog.939. PMID 14971006
- [Background] Baguley SD, Curnow JS, Morrison GD, Barron LF. Vaginal algometer: development and application of a device to monitor vaginal wall pressure pain threshold. Physiol Meas. 2003 Nov;24(4):833-6. doi: 10.1088/0967-3334/24/4/302. PMID 14658776
- [Background] Tu FF, Fitzgerald CM, Kuiken T, Farrell T, Norman Harden R. Vaginal pressure-pain thresholds: initial validation and reliability assessment in healthy women. Clin J Pain. 2008 Jan;24(1):45-50. doi: 10.1097/AJP.0b013e318156db13. PMID 18180636
- [Background] Tu FF, As-Sanie S, Steege JF. Musculoskeletal causes of chronic pelvic pain: a systematic review of diagnosis: part I. Obstet Gynecol Surv. 2005 Jun;60(6):379-85. doi: 10.1097/01.ogx.0000167831.83619.9f. PMID 15920438
- [Background] Nelson P, Apte G, Justiz R 3rd, Brismee JM, Dedrick G, Sizer PS Jr. Chronic female pelvic pain--part 2: differential diagnosis and management. Pain Pract. 2012 Feb;12(2):111-41. doi: 10.1111/j.1533-2500.2011.00492.x. Epub 2011 Jul 31. PMID 21801301
- [Background] Gyang A, Hartman M, Lamvu G. Musculoskeletal causes of chronic pelvic pain: what a gynecologist should know. Obstet Gynecol. 2013 Mar;121(3):645-650. doi: 10.1097/AOG.0b013e318283ffea. PMID 23635629
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] Bo K, Nygaard IE. Is Physical Activity Good or Bad for the Female Pelvic Floor? A Narrative Review. Sports Med. 2020 Mar;50(3):471-484. doi: 10.1007/s40279-019-01243-1. PMID 31820378
- [Background] Dehnavi ZM, Jafarnejad F, Kamali Z. The Effect of aerobic exercise on primary dysmenorrhea: A clinical trial study. J Educ Health Promot. 2018 Jan 10;7:3. doi: 10.4103/jehp.jehp_79_17. eCollection 2018. PMID 29417063
- [Background] Steege JF, Blumenthal JA. The effects of aerobic exercise on premenstrual symptoms in middle-aged women: a preliminary study. J Psychosom Res. 1993;37(2):127-33. doi: 10.1016/0022-3999(93)90079-u. PMID 8463989
- [Background] Awad E, Ahmed HAH, Yousef A, Abbas R. Efficacy of exercise on pelvic pain and posture associated with endometriosis: within subject design. J Phys Ther Sci. 2017 Dec;29(12):2112-2115. doi: 10.1589/jpts.29.2112. Epub 2017 Dec 7. PMID 29643586
- [Background] DeLong ER, DeLong DM, Clarke-Pearson DL. Comparing the areas under two or more correlated receiver operating characteristic curves: a nonparametric approach. Biometrics. 1988 Sep;44(3):837-45. PMID 3203132
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Dyck PJ, Boes CJ, Mulder D, Millikan C, Windebank AJ, Dyck PJ, Espinosa R. History of standard scoring, notation, and summation of neuromuscular signs. A current survey and recommendation. J Peripher Nerv Syst. 2005 Jun;10(2):158-73. doi: 10.1111/j.1085-9489.2005.0010206.x. PMID 15958127
- [Background] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Background] Hallett M. NINDS myotatic reflex scale. Neurology. 1993 Dec;43(12):2723. doi: 10.1212/wnl.43.12.2723. No abstract available. PMID 7802740
- [Background] Slieker-ten Hove MC, Pool-Goudzwaard AL, Eijkemans MJ, Steegers-Theunissen RP, Burger CW, Vierhout ME. Face validity and reliability of the first digital assessment scheme of pelvic floor muscle function conform the new standardized terminology of the International Continence Society. Neurourol Urodyn. 2009;28(4):295-300. doi: 10.1002/nau.20659. PMID 19090583
- [Background] Apte G, Nelson P, Brismee JM, Dedrick G, Justiz R 3rd, Sizer PS Jr. Chronic female pelvic pain--part 1: clinical pathoanatomy and examination of the pelvic region. Pain Pract. 2012 Feb;12(2):88-110. doi: 10.1111/j.1533-2500.2011.00465.x. Epub 2011 May 26. PMID 21615678
- [Background] Papoutsis D, Antonakou A. The Q-tip test of the vulva as a diagnostic aid for vulvodynia: sensitivity, specificity and predictive values. J Psychosom Obstet Gynaecol. 2019 Jun;40(2):90. doi: 10.1080/0167482X.2017.1415882. Epub 2017 Dec 19. No abstract available. PMID 29256294